CLINICAL TRIAL: NCT06121804
Title: The Cost-effectiveness Analysis of Immunosuppressants to Postoperative Infection and Death in the Patients With Organ Transplantation
Brief Title: Immunosuppressants to Postoperative Infection and Death
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CS2-21134
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Organ Transplantation; Immunosuppressive Agents; Cohort Study
MeSH Terms: interventions — Immunosuppressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with organ transplantation: Patients who underwent SOTs between 2002 and 2013, specifically, kidney (ICD-9-CM code V42.0), liver (ICD-9-CM code V42.7), or lung (ICD-9-CM code V42.6) transplants.
  Interventions: Drug: Immunosuppressive Agents
- Patients without organ transplantation: The general patients were enrolled as the comparison. We used propensity score matching (PSM) to establish a matched cohort.
  Interventions: Drug: Immunosuppressive Agents

INTERVENTIONS:
Drug: Immunosuppressive Agents — Prescribing immunosuppressive agents

SUMMARY:
The goal of this observational study is to explore the different immunosuppressive agents and related outcomes in organ transplantation patients in Taiwan. The main question it aims to answer is the risk of different immunosuppressive agents for infection and survival after transplant.

The study enrolled patients who underwent solid organ transplant (SOT), kidney (ICD-9-CM code V42.0), liver (ICD-9-CM code V42.7), or lung (ICD-9-CM code V42.6) transplants. We employed propensity score matching (PSM) to establish a matched cohort. The study will compare SOT patients and general patients to explore the risk of different immunosuppressive agents for infection and survival.

DETAILED DESCRIPTION:
This study used secondary data from the Longitudinal Health Insurance Database (LHID), a subset of the NHIRD provided by the Health and Welfare Data Science Center (HWDC) of the Ministry of Health and Welfare in Taiwan.

The HWDC encrypts personally identifying data to protect the privacy of beneficiaries. The database includes detailed clinical records from both the inpatient and outpatient claims of the beneficiaries of Taiwan's National Health Insurance program. This program has provided coverage for up to 99% of the country's population since 1995. The NHIRD can serve as a foundation for the procurement of real-world evidence to support clinical decisions and health-care policy-making.

Diagnostic data within the NHIRD from before 2016 and from 2016 or later are respectively coded using International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) and International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) codes.

The database was provided by the HWDC under license and so cannot be made freely available. Requests for access to these data should be made to HWDC (https://dep.mohw.gov.tw/dos/cp-5119-59201-113.html).

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent solid organ transplant (SOT)

Exclusion Criteria:

* Patients who received more than one SOT, had an infectious disease diagnosis before their SOT or had incomplete medical information in the database.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The present study enrolled patients who underwent SOTs between 2002 and 2013, specifically, kidney (ICD-9-CM code V42.0), liver (ICD-9-CM code V42.7), or lung (ICD-9-CM code V42.6) transplants. Patients were excluded from our study if they received more than one SOT, had an infectious disease diagnosis before their SOT, or had incomplete medical information in the NHIRD.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative infection | From the date of underwent SOTs until the date of incident infection or date of death from any cause, whichever came first, assessed up to 5 years.
  Postoperative infection contains Pneumocystis jiroveci pneumonia, cytomegalovirus disease, and Herpes simplex virus
Death | From the date of underwent SOTs until the date of death from any cause, assessed up to 5 years.
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ying Lee, PhD, Study Chair — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
The database used to support the findings of this study was provided by the Health and Welfare Data Science Center, Ministry of Health and Welfare (HWDC, MOHW) Taiwan under license and so cannot be made freely available. Requests for access to these data should be made to HWDC (https://dep.mohw.gov.tw/dos/np-2497-113.html).

REFERENCES:
- See also: The Health and Welfare Data Science Center, Ministry of Health and Welfare Taiwan — https://dep.mohw.gov.tw/DOS/cp-5119-59201-113.html